CLINICAL TRIAL: NCT00237276
Title: Evaluation of Effect of Colonoscopist Experience and Addition of of Mucosal Enhancement Techniques on Detection of Colonic Polyps When Viewing Videotaped Colonoscopic Withdrawals
Brief Title: Experience and Enhancement: Improving Colonoscopic Polyp Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 05/CL05/70
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Polyps
Keywords: colonoscopy, chromoendoscopy, autoflurescence, narrow band imaging, high definition endoscopy, colorectal cancer, colitis, polyp, DALM, adenoma, video
MeSH Terms: conditions — Polyps; Colorectal Neoplasms; Colitis; Adenoma | interventions — Colonoscopy

INTERVENTIONS:
Procedure: colonoscopy

SUMMARY:
The study looks at 2 hypotheses in 2 patient groups:

1. Are more experienced endoscopists better at detecting subtle lesions (polyps) on the lining of the colon (large bowel) than less experienced endoscopists?
2. Do existing and new techniques that can highlight lesions on the lining of the bowel improve endoscopists ability to spot them? This will be tested using video footage of endoscopies from 2 patient groups: those with a normal colon linig and those with colitis (bowel lining inflamation)

DETAILED DESCRIPTION:
Colorectal cancer is the second commonest cause of cancer death. In a majority of cases it is preceeded by a precancerous lesion called an adenoma (commonly known as polyp). Patients with colitis are at specially high risk of colorectal cancer which is estimated to be 18% at 30 years of disease. Detection and removal of adenomas at colonoscopy has been shown to reduce the death rate from colorectal cancer. However, despite meticulous examination there is a "miss rate" for adenomas at colonoscopy with ranges from 6-15% in back-to-back colonoscopy studies. The nature of the polyps which as well as being pedunculated (cherry like) can be flat or depressed making them difficult to see and may also contribute to the "miss rate".

The factors that affect whether an endoscopist sees a polyp are not well studied. Polyp detection rates vary widely, even amongst experts. Endoscopist experience is assumed to improve polyp detection rates; however in one study the least experienced endoscopists found the most polyps. Techniques that highlight lesions advanced in recent years. Chromoendoscopy, spraying dye on the bowel lining, has been shown to help pick up more pre-cancerous polyp in one of three studies in normal patients and seems definitely helpful in colitis. Autofluorescence endoscopy and narrow band imaging use light filters to produce a false colour image of the bowel lining where polyps stand out. These techniques have been used with some success in the oesophagus and stomach but little work is available for the colon. High definition endoscopy produces very clear images and may also help in polyp detection.

This study aims to collect videos of colonoscopy when the colonoscope is being removed. This is the main time when polyps are looked for. Some videos will have subtle polyps. The study will re-examine and re-video these areas using one of the techniques which may make polyps stand out better. The aim is to get videos of polyps with and without each of the techniques to highlight the lesions in both normal colon and colitis. These videos will then be shown to endoscopist of differing experience to test if their ability to spot the lesions depends on experience and to see if techniques to make lesions stand out help them see lesions more easily.

ELIGIBILITY:
Inclusion Criteria:

* Patients: over 18 years of age, with clinical indication for colonoscopy who are considered by the endoscopist to be fit for the procedure
* Endoscopists who have started colonoscopy training on a recognised training rotation. Consultants who perform colonoscopy regularly

Exclusion Criteria:

* patients under 18 years, patients with previous colorectal surgery or known familial polyposis, patients unable to give informed consent, pregnant patients, patients for whom coloscope insertion was difficult or uncomfortable, patients whose colon is not sufficiently cleared of stool, those unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
The difference in adenoma detection rate on video between consultants endoscopist vs. trainee endoscopists who have performed more than 200 endoscopies vs. trainee endospopists who have performed less than 200 endoscopies

SECONDARY OUTCOMES:
For each technique:
differences in adenoma detection rate between endoscopist of varying abilities with and without techniques to highlight polyps. Differences in adenoma detection rate in terms of esperience.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saunders, MD, FRCP, Principal Investigator — London North West Healthcare NHS Trust
Locations (1):
- North West London Hospitals NHS Trust - St Mark's Hospital, London, United Kingdom